CLINICAL TRIAL: NCT07378631
Title: Association Between Clinical Subtypes and Prognosis in Radiation Rectal Injury: A Prospective, Observational Study
Brief Title: Association Between Clinical Subtypes and Prognosis in Radiation Rectal Injury
Status: Recruiting | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: CRP202501
Record Dates: First submitted 2025-11-18; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Radiotherapy; Radiation Proctitis
Keywords: radiotherapy; radiation proctitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic radiation proctitis: Patients diagnosed with chronic radiation proctitis

SUMMARY:
This is a prospective, observational study aimed at exploring the associations between the clinical subtypes of radiation rectal injury and prognosis. The study is planed to commence in November 2025 and prospectively observe 150 patients. During the study period, researchers will not intervene in clinical treatment decisions but will only collect patient clinical information, intestinal endoscopy/imaging/pathological data, test results, and follow-up data. The study results will fill the evidence gap in this field, advance the diagnosis and treatment of radiation-induced rectal injury, and provide scientific support for improving the prognosis of similar patients.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years;
2. Diagnosed with radiation rectal injury.

Exclusion Criteria:

1. Ongoing cancer therapy;
2. Tumor recurrence or metastasis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of prospectively recruited adult patients clinically diagnosed with radiation rectal injury. Participants will be selected from the patient cohort at the Sixth Affiliated Hospital of Sun Yat-sen University. The inclusion criteria are: age between 18 and 80 years, and a clinical confirmation of radiation rectal injury. Patients who are currently undergoing cancer therapy or who have experienced tumor recurrence or metastasis are excluded. This study will be conducted in accordance with the Declaration of Helsinki and has been approved by the hospital's Ethics Committee. Written informed consent will be obtained from all participants prior to their enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Association between Clinical Classification and Clinical Outcomes | 6 months
  To investigate the association between clinical subtypes and outcomes, the primary outcome was assessed as complete remission of their primary symptom, while the measure was identified as the remission rate.

SECONDARY OUTCOMES:
Predictive Accuracy of Endoscopic Characteristics for Clinical Subtyping | 6 months
  Using prospectively collected endoscopic data, the investigators will assess the association between specific endoscopic features and the data-driven clinical subtypes. The predictive accuracy will be quantitatively measured using metrics including sensitivity and specificity. The results aim to determine whether endoscopic findings can serve as reliable indicators for subtype identification.
Predictive Accuracy of Imaging Evaluation for Clinical Subtyping | 6 months
  Using prospectively collected endoscopic data, the investigators will assess the association between features of MRI/CT and the data-driven clinical subtypes. The predictive accuracy will be quantitatively measured using metrics including sensitivity and specificity. The results aim to determine whether endoscopic findings can serve as reliable indicators for subtype identification.

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China